CLINICAL TRIAL: NCT04997213
Title: Effects of Classical Balance-Coordination Exercises and Static Posturography Device Assisted Feedback Exercises on Fall Risk and Balance-Coordination Parameters in Parkinson Disease
Brief Title: Biofeedback Balance Exercises in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif yaksi, Medical Doctor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-FTR-EY-05
Record Dates: First submitted 2021-07-28; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease; Balance; Distorted
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: We have two groups. First group received biofeedback exercise and conventional exercise group, second group received only conventional exercise treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Biofeedback system is a center of pressure-controlled video game-based exercise system designed for patients with neurological and orthopedic diseases and provides balance training using auditory, visual, and pressure biofeedback. The system contains several games, each designed to focus on a different component of balance. Biofeedback is provided by means of a monitor in front of the patient. The balance exercises program involved a total of 18 sessions, each lasting 20 min, three times a week for six weeks, and were individually tailored based on the patient's tolerance and current motor and sensorial capacities. All patients performed conventional exercises.
  Interventions: Other: Biofeedback exercises; Other: Conventional Exercises
- Control group (Active Comparator): Classic balance exercises were performed (two-leg stance, semi-tandem stance, tandem stance, standing on one leg, tandem walking, turning completely around, heel-to-toe stance, and standing with the eyes closed). Patients with balance disorder first were commenced balance training in a seated position before progressing to standing exercises, to the extent that these could be tolerable.
  Interventions: Other: Conventional Exercises

INTERVENTIONS:
Other: Biofeedback exercises — Biofeedback system is a center of pressure-controlled video game-based exercise system designed for patients with neurological and orthopedic diseases and provides balance training using auditory, visual, and pressure biofeedback. The system contains several games, each designed to focus on a different component of balance. Biofeedback is provided by means of a monitor in front of the patient. The balance exercises program was involved a total of 18 sessions, each lasting 20 min, three times a week for six weeks, and was individually tailored based on the patient's tolerance and current motor and sensorial capacities. All patients performed conventional exercises.
  Arms: Interventional group
Other: Conventional Exercises — Classic balance exercises were performed (two-leg stance, semi-tandem stance, tandem stance, standing on one leg, tandem walking, turning completely around, heel-to-toe stance, and standing with the eyes closed). Patients with balance disorder first could be commenced balance training in a seated position before progressing to standing exercises, to the extent that these could be tolerable.

SUMMARY:
The aim of this study was to evaluate the effectiveness of static posturography-assisted biofeedback exercises in PD-related balance disorder.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a chronic, progressive, degenerative movement disorder, the incidence of which increases with age, characterized by motor and non-motor findings. Cardinal motor findings such as bradykinesia, rigidity, rest tremor, postural instability, and gait dysfunction and secondary motor symptoms additional to these such as dysarthria, and associated movements in the arms may be seen throughout the course of the disease. Progressive loss of dopaminergic neurons occurs in the basal ganglia, together with a decrease in the speed and angle of movement. Loss of postural reflexes causes balance disturbance findings such as impaired postural control, rigidity in the extremities, and akinesia.Falls, decreased mobility, disability and quality of life impairment occur as a result of balance disorder. Higher rates of falls or fall-related fractures have been reported in PD compared to the non-PD elderly population.There are several exercise applications aimed at balance improving strategies in PD. Strengthening exercises combined with conventional balance exercises, treadmill walking training, tai chi, and biofeedback have been shown to improve gait and and balance control in PD. Various publications have shown that biofeedback therapy in elderly individuals and in healthy individuals with postural disorder exhibits positive effects on balance by enhancing postural stability and reducing body tremor. The basic aim of this study was to investigate the effects of static posturography-assisted visual and auditory biofeedback therapy on balance and the risk of falls in PD. In addition, the study was intended to determine the effects of balance training on the individual's daily living activities, perceived safety level, and emotional state.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease,
* Age 40 - 85

Exclusion Criteria:

* Presence of systemic or neurological disease capable of causing balance disorder,
* Postural hypotension,
* Presence of cardiovascular or musculoskeletal system disease capable of affecting locomotion,
* Presence of advanced dementia or mental disability

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
The Hoehn and Yahr Scale | Baseline
  All patients in this study were classified based on the Hoehn and Yahr scale prior to treatment. This scale is widely used for classifying PD into five stages. It permits objective evaluation of the progression of the disease, from Stage 0 (no disease symptoms) to Stage 5 (the patient is confined to a wheelchair or bed).
The Movement Disorder Society Unified Parkinson's Disease rating Scale | Baseline
  This is an extensive scale employed for the clinical evaluation of severity of PD. It consists of four sections including non-motor findings, motor problems, motor findings, and treatment complications. Fourteen motor findings (0 - no finding, or normal, 4- severe finding) in the second section of the scale and comprising the motor problems part were evaluated before treatment in this study.
The Movement Disorder Society Unified Parkinson's Disease rating Scale | 6 weeks
  This is an extensive scale employed for the clinical evaluation of severity of PD. It consists of four sections including non-motor findings, motor problems, motor findings, and treatment complications. Fourteen motor findings (0 - no finding, or normal, 4- severe finding) in the second section of the scale and comprising the motor problems part were evaluated before treatment in this study.
Tinetti Balance and Gait Assessment | Baseline
  This scale consists of two sections assessing gait and balance. The first nine questions concern balance, and the following seven concern gait. The total possible score is 28, consisting of 12 for the gait scale and 16 for the balance scale
Tinetti Balance and Gait Assessment | 6 weeks
  This scale consists of two sections assessing gait and balance. The first nine questions concern balance, and the following seven concern gait. The total possible score is 28, consisting of 12 for the gait scale and 16 for the balance scale
Berg Balance Scale | Baseline
  This scale consists of 14 sections and measures the ability to maintain balance during voluntary movements and postural changes in the trunk and extremities. Scoring is between 0 and 4 (0: unable to complete the task, 4: normal performance). The highest possible score is 56. Scores of 0-20 indicate balance disorder, scores of 21-40 indicate acceptable balance, and scores of 41-56 indicate good balance
Berg Balance Scale | 6 weeks
  This scale consists of 14 sections and measures the ability to maintain balance during voluntary movements and postural changes in the trunk and extremities. Scoring is between 0 and 4 (0: unable to complete the task, 4: normal performance). The highest possible score is 56. Scores of 0-20 indicate balance disorder, scores of 21-40 indicate acceptable balance, and scores of 41-56 indicate good balance
Timed Up and Go Test | Baseline
  TUG evaluation was performed before and after treatment. In this test, the subject is asked to stand up from a chair, walk 3 meters, turn around, walk back to the chair and sit back down, and the time taken to perform this task is recorded in seconds.
Timed Up and Go Test | 6 weeks
  TUG evaluation was performed before and after treatment. In this test, the subject is asked to stand up from a chair, walk 3 meters, turn around, walk back to the chair and sit back down, and the time taken to perform this task is recorded in seconds.

SECONDARY OUTCOMES:
Tandem Stance Test | Baseline
  Tandem stance is a clinical measurement used to assess postural stability and standing balance in a heel-to-toe position on a narrow base of support with a temporal measurement. The individual's ability to maintain static balance is recorded in seconds
Tandem Stance Test | 6 weeks
  Tandem stance is a clinical measurement used to assess postural stability and standing balance in a heel-to-toe position on a narrow base of support with a temporal measurement. The individual's ability to maintain static balance is recorded in seconds
Health Assessment Questionnaire | Baseline
  This questionnaire consists of eight questions designed to assess the effects of individuals' health status on daily living. Day-to-day activities such as dressing, hygiene, eating, and walking are assessed, and high scores indicate poor health status.
Health Assessment Questionnaire | 6 weeks
  This questionnaire consists of eight questions designed to assess the effects of individuals' health status on daily living. Day-to-day activities such as dressing, hygiene, eating, and walking are assessed, and high scores indicate poor health status.
Beck Depression Inventory | Baseline
  The BDI is used to evaluate physical, emotional, and cognitive symptoms encountered in depression, such as hopelessness, irritability, guilt, fatigue, and weight loss. Scoring is performed from absence of symptoms to severe symptoms. Total scores range between 0 (no depression) and 63 (severe depression).
Beck Depression Inventory | 6 weeks
  The BDI is used to evaluate physical, emotional, and cognitive symptoms encountered in depression, such as hopelessness, irritability, guilt, fatigue, and weight loss. Scoring is performed from absence of symptoms to severe symptoms. Total scores range between 0 (no depression) and 63 (severe depression).

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yakşi, MD, Principal Investigator — Abant İzzet Baysal University Medical Faculty
Locations (1):
- Elif Yakşi, Bolu, Turkey (Türkiye)